CLINICAL TRIAL: NCT04604938
Title: The Role of the Renin-angiotensin System in Reward Reinforcement Learning
Brief Title: The Effects of Losartan on Reward Reinforcement Learning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-75
Record Dates: First submitted 2020-10-09; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Healthy
Keywords: Losartan; Reward reinforcement learning
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan group (Experimental): Drug: Losartan
  Interventions: Drug: Losartan
- Placebo group (Placebo Comparator): Drug: Placebo Oral Tablet
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Losartan — administration of losartan (50 mg) (oral)
  Other Names: Cozaar Oral Tablet
  Arms: Losartan group
Drug: Placebo oral tablet — administration of placebo (oral)
  Arms: Placebo group

SUMMARY:
This study aims to investigate whether a single dose of losartan (50 mg) can affect learning from positive and negative outcomes and its related neural mechanisms.

DETAILED DESCRIPTION:
Emerging evidence suggests that the renin-angiotensin system can impact dopamine (DA) transmission and its modulatory role in reward processing. For instance, recent animal models have found that the angiotensin antagonist losartan reduces rewarding effects of methamphetamine and nicotine by modulating DA release in the striatum.The present study thus will investigate losartan effects on reward reinforcement learning and the underlying neural mechanisms. In a double-blind, between-subject, placebo-controlled design, 60 healthy male subjects will be randomly assigned to receive single-dose losartan (50 mg) or placebo, 90 minutes before performing a probabilistic reinforcement learning task during fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders
* Right-handedness
* Normal or corrected-normal version

Exclusion Criteria:

* History of head injury
* Medical or psychiatric illness
* Hypertension
* General cardio-vascular alteration or diseases
* Allergy against medications
* Visual or motor impairments
* Claustrophobia
* Drug addiction
* Nicotine dependence
* FMRI contradictions

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
BOLD-level activity as assessed by fMRI during the learning phase | 90 minutes to 110 minutes after treatment
  During the paradigm subjects will learn the reward properties of stimuli via the presentation of trial-wise feedback. The neural activation during the prediction of positive and negative outcome feedback will be assessed by functional magnetic resonance imaging (fMRI), particularly in prefrontal and subcortical regions. The effects of treatment will be determined by comparing the losartan- and placebo-treated groups.
BOLD-level activity as assessed by fMRI during the learning transfer phase | 111 minutes to 120 minutes after treatment
  Following the initial learning phase subjects learning transfer will be examined by asking subjects to choose between stimuli with high versus low reward probabilities. The neural activation during correct responses will be assessed by functional magnetic resonance imaging (fMRI), particularly in prefrontal and subcortical regions. The effects of treatment will be determined by comparing the losartan- and placebo-treated groups.

SECONDARY OUTCOMES:
Choice accuracy for the stimulus with the high reward probability during the learning phase | 90 minutes to 110 minutes after treatment
  During the learning phase accuracies (in percent) for choosing the stimulus with the highest reward probability will be computed. Effects of treatment on choice accuracy in the probabilistic learning task will be examined by comparing accuracies (percent) between the losartan- and placebo-treated group.
Learning rate for positive and negative outcomes | 90 minutes to 110 minutes after treatment
  The learning rate will be determined by performing computational modelling. The learning rate index for positive and negative outcomes during the learning phase will be compared between the losartan- and placebo-treated group.
Choice accuracy during the learning transfer phase | 111 minutes to 120 minutes after treatment
  Following the initial learning phase subjects learning transfer will be examined by asking subjects to choose between stimuli with high versus low reward probabilities. For the transfer phase the choice accuracy for selecting stimuli with the highest reward probability and avoiding stimuli with the lowest reward probability will be computed. The effects of treatment will be determined by comparing the accuracy between the losartan- and placebo-treated groups.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu T, Zhou X, Kanen JW, Wang L, Li J, Chen Z, Zhang R, Jiao G, Zhou F, Zhao W, Yao S, Becker B. Angiotensin blockade enhances motivational reward learning via enhancing striatal prediction error signaling and frontostriatal communication. Mol Psychiatry. 2023 Apr;28(4):1692-1702. doi: 10.1038/s41380-023-02001-6. Epub 2023 Feb 21. PMID 36810437